CLINICAL TRIAL: NCT05497570
Title: Does Intra-articular Injection of Tenoxicam After Arthrocentesis Heal Outcomes of Temporomandibular Joint Osteoarthritis? A Randomized Clinical Trial
Brief Title: Injection of Tenoxicam Versus Arthrocentesis Alone in the Treatment of Temporomandibular Joint Osteoarthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Zeynep Bayramoglu, Assistant Professor, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3525
Record Dates: First submitted 2022-08-05; First posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Arthrocentesis
MeSH Terms: interventions — Arthrocentesis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenoxicam (Active Comparator): The Tenoxicam group (n:16) received both arthrocentesis and a 2-ml injection of tenoxicam (Oksamen-L, Mustafa Nevzat İlaç Sanayi, Istanbul, Turkey) to the temporomandibular joint.
  Interventions: Drug: Tenoxicam Injectable Product
- Control (Active Comparator): Only arthrocentesis was given to patients in the control group
  Interventions: Drug: Tenoxicam Injectable Product

INTERVENTIONS:
Drug: Tenoxicam Injectable Product — After arthrocentesis procedure, 2-ml injection of tenoxicam (Oksamen-L, Mustafa Nevzat İlaç Sanayi, Istanbul, Turkey) to the temporomandibular joint
  Other Names: Arthrocentesis

SUMMARY:
The aim of the study is to examine the effectiveness of arthrocentesis plus tenoxicam injection and to compare it with arthrocentesis alone in patients with TMJ-OA.

Thirty patients with TMJ-OA who were treated randomly with either arthrocentesis plus tenoxicam injection (TX group) or arthrocentesis alone (control group) were examined. Maximum mouth opening (MMO), visual analog scale (VAS) pain values, and joint sounds were the outcome variables, which were evaluated at pre-treatment and at 1, 4, 12, and 24 weeks after treatment.

DETAILED DESCRIPTION:
Temporomandibular joint osteoarthritis (TMJ-OA) is a very painful disease that disrupts the patient's comfort of life. Arthrocentesis alone or in combination with intraarticular injections is highly effective in the treatment of TMJ-OA. It reduces pain, increases mouth opening, and improves jaw movements. In intra-articular injections, hyaluronic acid, platelet-rich plasma, corticosteroids, and non-steroidal anti-inflammatory drugs (NSAIDS) are used. Tenoxicam is an NSAID that is used systemically or locally in joint diseases such as acute or chronic inflammatory rheumatoid arthritis and osteoarthritis. It has been reported that its long-lasting analgesic effect and anti-inflammatory effect are higher in intra-articular administration than in oral and intravenous administrations , to our knowledge, there has been no such study analysing the effectiveness of intra-articular application of tenoxicam in patients with TMJ-OA. The aim of the study is to examine the effectiveness of arthrocentesis plus tenoxicam injection and to compare it with arthrocentesis alone in patients with TMJ-OA.

Thirty patients with TMJ-OA who were treated randomly with either arthrocentesis plus tenoxicam injection (TX group) or arthrocentesis alone (control group) were examined. Maximum mouth opening (MMO), visual analog scale (VAS) pain values, and joint sounds were the outcome variables, which were evaluated at pre-treatment and at 1, 4, 12, and 24 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and radiological diagnosis of TMJ-OA
* 18 years of age and older
* Sufficient clinical data at baseline and follow-up.

Exclusion Criteria:

* Uncontrolled systemic disease
* Neurological disease
* Previous TMJ surgery
* Malignant disease in the head and neck region

Ages: 22 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2019-05-03 (Actual); Primary Completion 2021-11-07 (Actual); Study Completion 2022-04-21 (Actual)

PRIMARY OUTCOMES:
Pain on Tmj (Visual analog scale(VAS) was used.) | Change from baseline pain on TMJ at six months
  Pain scores of Temporomandibular joint on a visual analog scale.To measure the VAS value, a 10-cm-long numbered line was created. The patient chose a point on the line, the corresponding value was measured with a ruler, and a score was given. 0 means no pain and best outcome score; 10 means maximum pain and the worst score.
Maximum Mouth Opening(MMO) (A ruler was used) | Change from baseline maximum mouth opening at six months
  MMO was gaged with a ruler between the incisal edges of the maxillar and mandibular central incisors when the patient open the mouth maximum. The score was written in mm.
Joint sounds (Visual analog scale was used to measure.) | Change from baseline joint sounds at six months
  Temporomandibular joint sounds was measured with Visual analog scale (VAS).To measure the VAS value, a 10-cm-long numbered line was created. The patient chose a point on the line, the corresponding value was measured with a ruler, and a score was given. 0 means no sounds and best outcome score; 10 means maximum sound and the worst score.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Bayramoglu, Study Director — Ataturk University
Locations (1):
- Ataturk University, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bayramoglu Z, Yavuz GY, Keskinruzgar A, Koparal M, Kaya GS. Does intra-articular injection of tenoxicam after arthrocentesis heal outcomes of temporomandibular joint osteoarthritis? A randomized clinical trial. BMC Oral Health. 2023 Mar 8;23(1):131. doi: 10.1186/s12903-023-02852-z. PMID 36890529